CLINICAL TRIAL: NCT05900934
Title: The Effects of Myofascial Release in Combined With Task-oriented Circuit Training on Balance and Gait in People With Parkinson's Disease
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Kutay Kaslı, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KA-22060
Record Dates: First submitted 2023-05-23; First posted 2023-06-13 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Parkinson Disease; Myofascial Release; Exercise Therapy; Movement Disorders
Keywords: myofascial releasing; gait; balance
MeSH Terms: conditions — Parkinson Disease; Movement Disorders | interventions — Myofascial Release Therapy

STUDY DESIGN:
Intervention Model Description: Arm 1: Myofascial Releasing Group Arm 2: Sham Myofascial Releasing Group
Who Masked: Participant, Outcomes Assessor
Masking Description: A double-blind, assessor-blinded and patient-blinded, randomized controlled study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myofascial Releasing Group (Active Comparator): The intensity of application is important for foam rollers. For intensity, the intensity of the pressure will be determined by a subjective 7/10 target numeric rating scale rating (0 representing no discomfort and 10 representing maximum discomfort) and applied at the end of each session.
  Interventions: Other: Myofascial Releasing Group
- Sham Myofascial Releasing Group (Sham Comparator): In the sham group, similar to the literature, the intensity will be applied with foam rollers in accordance with the 0/10 numerical rating scale, to the same application areas, for the same duration and with the same rest intervals.
  Interventions: Other: Sham Myofascial Releasing Group

INTERVENTIONS:
Other: Myofascial Releasing Group — Using a subjective 7/10 target numeric rating scale rating (0 representing no discomfort and 10 representing maximum discomfort), the intensity of foam roller application can be determined. This intensity defines an application intensity that is mildly painful for the participant and appropriate according to previous literature.
  Other Names: Myofascial Release
  Arms: Myofascial Releasing Group
Other: Sham Myofascial Releasing Group — The severity of the application is not felt at all according to the numerical rating scale of 0/10.
  Other Names: Sham Myofascial Release
  Arms: Sham Myofascial Releasing Group

SUMMARY:
In this study, the investigators plan to have Parkinson's patients perform exercises according to the task-oriented training method. Since recent studies have suggested that task-oriented training should be organized as a series of workstations that allow for more intensive practice, each of them has a program content implemented in the form of a station. The program will be implemented in 11 different stations with 3 minutes and a 1-minute break at each station, 3 days a week for 8 weeks under the supervision and guidance of a physiotherapist. The task-oriented training program will be carried out by applying the above-mentioned exercises in the form of stations sequentially within a certain period of time. For all exercises, the intensity perceived by the individuals will be ensured to be 12-15 points of perceived exertion according to the Borg Perceived Exertion Scale. In this way, the exercise program can be easily individualized according to the participant's pain, complaints, and functional status. In the study, after the task-oriented approach, foam roller application and myofascial release will be applied at the end of each session.

Foam roller application; C7-T1 and posterior neck region, thoracic spine, lumbar spine, and right and left sides of the thoracolumbar spine will be applied with a foam roller, which is a myofascial release device, in each session. Each application area will be applied in 3 sets of 60 seconds of application and 30 seconds of rest. The intensity of the pressure for the intensity of the application will be subjectively controlled with a target numeric rating scale rating of 7/10 (0 represents no discomfort and 10 represents maximum discomfort). In the sham group, similar to the literature, the intensity of the application will be applied in accordance with the 0/10 numeric rating scale, at the same application sites, for the same duration and the same rest intervals.

Within the scope of this study, participants gait, balance, rotation time, range of motion, level of achievement of the treatment goal, quality of life and trunk impairment will be evaluated at the beginning of the study and at the end of 8 weeks.

DETAILED DESCRIPTION:
Participants who meet the inclusion criteria will be randomly divided into 2 groups as 'PH-Myofascial Release Group' and 'PH-Sham Myofascial Release Group' as the control arm by closed envelope method. In this randomized controlled study, the noninvasive application will be performed with Foam rollers for the same duration, same muscle area, same set intervals and same number of sets in both groups. The intensity of the applications will be different for the research arm (PH-Myofascial Relaxation Group) for the C7-T1 spine and posterior neck region of the body, thoracic spine, lumbar spine, thoracolumbar spine right and left sides of the body according to the Numeric Pain Scale 7/10 and for the control arm (PH- Sham Myofascial Relaxation Group) 0/10 intensity on the same scale will be applied as applied in the literature. After the exercise application called task-oriented training protocol is applied to both groups, foam roller application time will be applied to each application area as 3 sets of 60 s applications and 30 s rest. The application will be performed 3 days a week for 8 weeks under the supervision of a physiotherapist. Task-oriented training; It has a program content consisting of coming from sitting to standing, standing, get up and walk exercise, walking exercise on the inclined ground, step exercise, slalom exercise, stair exercise, touching different points in the mirror exercise, reaching exercise, boxing exercise, balance exercise on moving ground, mat exercise, writing, eating exercise, each of which is applied in the form of a station. Since the limitation in the trunk in Parkinson's disease may also be caused by non-neural structures, it is curious to evaluate the effects of myofascial release. The effects of myofascial release when applied in combination with a task-oriented exercise approach compared to the sham application have not yet been shown on basic motor parameters such as balance and gait in neurological diseases. Based on these premises, the aim of the study was to evaluate the effects of foam roller application in patients with Parkinson's disease when applied in combination with a rehabilitation program.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with "Parkinson's Disease" by a specialist physician,
* In a stable period in terms of motor fluctuations and drug treatment
* Severity of the disease (1-3 according to Hoehn & Yahr) staging
* No other neurological disease
* Cognitive status of 24 and above according to the Mini-Mental State Evaluation (MMSE) test
* No change in Parkinson's disease-related medications or doses during the study
* Volunteering to participate in the study and giving written informed consent

Exclusion Criteria:

* Hearing and visual impairment, orthopedic, cardiopulmonary and additional neurological diseases that prevent participation in exercises
* Lack of independent ambulation
* Using a brain pacemaker for Parkinson's disease
* Continue with another rehabilitation program
* The occurrence of any health problem during the assessments and exercise training
* Failure to attend three consecutive sessions and a total of five sessions during the 24-session treatment

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2024-06-15 (Estimated); Study Completion 2024-09-15 (Estimated)

PRIMARY OUTCOMES:
GAITRite® gait system | Eight week
  Evaluation of time-distance characteristics of gait

SECONDARY OUTCOMES:
Berg Balance Scale | Eight week
  It is used to assess balance in the elderly and to determine the risk of falls. In the test consisting of 14 items, 0 points are given when the individual cannot perform the activity at all, and 4 points are given when the individual completes the activity independently. The maximum total score is 56. 0 to 20 points indicate a high risk of falling and impaired balance; 21 to 40 points indicate a moderate risk of falling and acceptable balance. 41 and above indicates good balance and minimal fall risk.
Posturographic assessment | Eight week
  With the Bertec Balance Check ScreenerTM force platform system (BP5050, Bertec Co., Columbus, OH, USA), stability limits in 4 different directions (front, back, right, left) will be evaluated on hard ground with eyes open and hard ground with eyes closed and also on soft ground.
The Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale | Eight week
  It evaluates Parkinson's disease in terms of mental and emotional state, motor examination, activities of daily living and treatment complications. A higher score indicates worse disease severity.
Roll-over test | Eight week
  Both 360-degree turns are timed with a stopwatch.
Range of Motion Assessment | Baseline- End of the eight week
  Neck flexion, extension, rotation, lateral flexion, trunk flexion, extension, rotation, lateral flexion and ankle dorsiflexion ROM will be measured.
Timed-up and go test | Eight week
  The timed up-and-go test will be measured without dual-task conditions and with cognitive and motor dual-task conditions.
Goal Attainment Scale | Eight week
  After the treatment, it allows patients to score the extent to which their individual goals have been achieved. GAS gives individuals the ability to construct their own outcome measures; this is in contrast to measures that are based on a standard set of tasks. Scoring, however, is performed in a standardised way which in turn allows for statistical analysis.GAS comprises of goals divided into a 5-point scale from -2 to +2.
The Parkinson's disease questionnaire-8 | Eight week
  It is an 8-question short form of the 39-item Parkinson's Disease Questionnaire developed specifically for the assessment of quality of life in Parkinson's disease.
Trunk impairment scale | Eight week
  It assesses static and dynamic sitting balance and trunk coordination. This scale comprises 17 items. The total score ranges from a minimum of 0 to a maximum 23 points, higher scores indicate better performance.
Body-Mass Index | Eight week
  Participants weight and height will be assessed by investigators and BMI will calculated by investigators.

CONTACTS AND LOCATIONS:
Overall Officials: Yahya Doğan, Dr, Principal Investigator — Hacettepe University; Muhammed Kılınç, Prof, Study Chair — Hacettepe University; Mert Doğan, PhD, Study Chair — Akdeniz University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kasli K, Dogan M, Ozal C, Dogan Y, Kilinc M, Aksu Yildirim S. The Effects of Foam Rolling after Task-Oriented Circuit Training on Gait, Balance, and Range of Motion in Parkinson's Disease: A Randomised Controlled Trial. Neurodegener Dis. 2025 Dec 26:1-12. doi: 10.1159/000550230. Online ahead of print. PMID 41452784
- [Derived] Kasli K, Dogan M, Ozal C, Dogan Y, Kilinc M, Aksu Yildirim S. The effects of myofascial release in combined with task-oriented circuit training on balance in people with Parkinson's disease: a randomized pilot trial. Neurol Res. 2024 Sep;46(9):848-858. doi: 10.1080/01616412.2024.2360860. Epub 2024 May 31. PMID 38818769